CLINICAL TRIAL: NCT06715566
Title: More Steps Towards an Active Life - ActForStroke
Brief Title: More Steps Towards an Active Life After Stroke - ActForStroke
Acronym: ActForStroke
Status: Not yet recruiting | Phase: Not Applicable | Type: Interventional
Sponsor: University of Aarhus (Other)
Collaborators: Regional Hospital Hammel Neurorehabilitation Centre (Unknown); University College Nordjylland (Unknown)
Responsible Party: Sponsor
Allocation: Non-Randomized | Model: Parallel | Masking: Single | Purpose: Treatment
Other Study IDs: ActForStroke; R260-A5988 Act for stroke (Other Grant/Funding Number: Danske Regioner - Forebyggelsespuljen)
Record Dates: First submitted 2024-11-18; First posted 2024-12-04 (Actual); Last update posted 2024-12-04 (Actual); Status verified 2024-11

CONDITIONS: Stroke Not Otherwise Specified
Keywords: stroke; activity; gait; training; coaching
MeSH Terms: conditions — Stroke; Motor Activity | interventions — Standard of Care

STUDY DESIGN:
Intervention Model Description: Parallel group quasi-experimental design
Who Masked: Outcomes Assessor
Oversight: Data Monitoring Committee: No | FDA-regulated Drug: No | FDA-regulated Device: No | US Export: No

ARMS (2):
- ActForStroke (Experimental): A combination of high-intensity gait training and coaching to encourage physical and social activity.
  Interventions: Behavioral: ActForStroke
- Standard care (Active Comparator): Standard care usually provided
  Interventions: Behavioral: Standard care

INTERVENTIONS:
Behavioral: ActForStroke — ActForStroke is a combination of 10 sessions high-intensity gait training and subsequent with up 7 coaching sessions until 1 year after stroke.
  Arms: ActForStroke
Behavioral: Standard care — Usual rehabilitation services
  Arms: Standard care

SUMMARY:
The main goal of this quasi-experimental study is to prevent the negative consequences of mobility impairments after stroke. These include recurrent strokes, general deconditioning, and overweight on the physical side, and dependency, isolation, caregiver strain, and reduced quality of life from a psycho-social perspective.

ActForStroke, a combination of high-intensity gait training and subsequent remote coaching and activity monitoring, will contribute to more steps, higher activity levels and increased participation. ActForStroke requires minimal extra resources and can easily be implemented within existing staffing levels.

The investigators want to examine if patients who participate in the ActForStroke intervention are more active one year after stroke.

Patients with stroke will either participate in a combined intervention of high-intensity gait training and subsequent coaching to facilitate physical and social activity or receive standard care.

DETAILED DESCRIPTION:
Stroke is worldwide the second most common cause of long-term disability. In Denmark, stroke affects around 12,000 people each year, and around 110,000 are living with the consequences of a stroke. One in five Danes over 25 will experience a stroke during their lifetime, and 30% of stroke victims are under 65 years old. These numbers imply not only a significant burden for the individual and their caregivers but also for society in general. The costs for treatment and care amount to 2.03 billion DKK annually, not including lost working capacity. People living with the consequences of a stroke are at a high risk of early death, recurrent strokes (around 10-26 % during the first years), and myocardial infarctions, aggravated by risk factors, such as diabetes and overweight, both from prior to stroke and after. A huge amount of evidence supports the preventive effect of physical activity in everybody, including those with stroke and comorbidities or other medical issues. To achieve a sufficient level of physical activity according to official recommendations (>30 min moderate activity per day plus 2 x 20 min vigorous activity per week) is challenging for almost everybody but can be especially challenging for people with stroke due to reduced mobility.

Gait after stroke Around two-thirds of those affected suffer from impaired gait function which limits their independence and participation in valued activities and compromises their physical fitness and psycho-social well-being. Recovery of walking early following neurologic injury is a primary goal of patients and their families. However, many walk at a slow pace and for limited distances. A majority of patients still suffer from reduced walking ability at discharge from the hospital. This can lead to a more homebound life with a reduction of social relations and a less active everyday life. Studies suggest that even small declines in gait speed from baseline (i.e., change of 0.1 m/s) are associated with significant increases in health care utilization (e.g., medical/surgical visits, hospitalization duration).

Inactivity after stroke is a consequence of walking impairment or just co-occurring with it, many people with stroke spend too much of their time sedentary and physically inactive. Studies indicate that people with stroke spend more time sedentary and in long uninterrupted sedentary bouts than age-matched healthy people. Interestingly, physical activity seems not to be directly related to their functional level. As inactivity is directly associated with increased cardiovascular risk, the risk for recurrent strokes increases.

ActForStroke With ActForStroke, the investigators want to address these challenges with the following combined interventions that are intended to start during inpatient rehabilitation and continue in municipality rehabilitation.

High-intensity gait training (HIGT) is based on substantial amounts of stepping practice at 70-85 % maximum heart rate. HIGT has been proven effective in other countries in enabling patients with stroke to achieve better gait and balance and, thus increasing their opportunities for an active and independent life. The effect could be maintained 1 year after stroke. Intensive gait training is now recommended by national guidelines for stroke rehabilitation in the US, UK, and Australia. HIGT is an approach that can be implemented within existing staffing levels and thus constitutes a viable long-term approach. However, it is usual practice in Denmark.

Encouraging an active lifestyle after discharge. While in-hospital rehabilitation is important, long-term efforts are needed to avoid deterioration of function. Underpinned by the behavior change theory, others, and own research, the investigators want to provide systematic and motivating coaching and activity monitoring to facilitate physical and social activity and to increase the likelihood that activity levels are maintained or extended and that physical activity becomes a daily routine. Moreover, the investigators want to contribute to the prevention or attenuation of the negative consequences of stroke resulting from an inactive, sedentary lifestyle.

In summary, inactivity and sedentary behavior after stroke is a substantial risk factor for recurrent strokes, other cardiovascular events, deterioration of function, and reduced health-related quality of life.

To achieve the overarching purpose of preventing negative effects of immobility caused by impaired gait function and sedentary behavior, the investigators aim to pursue 2 related objectives:

To achieve the best possible gait function during institutional rehabilitation and To maintain gait function and to achieve activity levels that are relevant as secondary prevention and satisfying and beneficial for the individual.

Methods 3.1. Design and settings This is a non-randomized control group study. It builds on an existing collaboration where one part of ActForStroke, HIGT, has already been introduced to therapists and first experiences have been made. The aim of the collaboration is to systematically examine the effect of ActForStroke and to provide a platform for knowledge sharing and the exchange of experiences. For the project, the collaboration has been complemented with other institutions (neurorehabilitation hospitals and municipality rehabilitation services) that have access to comparable patients or clients. Both quantitative and qualitative methods will be applied. Depending on the results, a larger randomized stepped-wedge design is planned.

The participating institutions reflect a variety of different settings and healthcare levels.

A. Intervention sites where ActForStroke is applied:

A1) In-hospital neurorehabilitation: Regionshospitalet Hammel Neurocenter (RHN) is a specialized hospital for the neurorehabilitation of acquired brain injuries. It has 110 beds and serves the entire region of Western Denmark.

Neuroenhed Nord is a regional specialized hospital for neurorehabilitation of acquired brain injuries. It has 52 beds and serves North Jutland.

and A2) Outpatient neurorehabilitation intervention sites: Aalborg municipality with 222.571 inhabitants, Thisted municipality with 43.160 inhabitants and, Jammerbugt municipality 38.500 inhabitants are municipalities of large, medium, and small sizes.

B. Control sites where standard care is applied B1) Neurorehabiliteringsafsnit NR, Svendborg, Neurologisk Afdeling N OUH, is a specialized neurorehabilitation hospital. It has 50 beds and serves the region of southern Denmark.

Neurocenter København, Department of brain and spinal cord injuries, is a specialiced hospital for the neurorehabiliation of acquired brain injuries and serves the region of Eastern Denmark, Greenland and the Faroe Islands. It was recently opened and has a total of 125 beds.

B2) Outpatient neurorehabilitation control sites consist of Vejle municipality with 121.616 inhabitants, Skive municipality with 45.069 inhabitants, and Favrskov with 49.408 inhabitants.

Participants from intervention sites will be compared to participants from control sites who are similar with regard to age, gender, severity of stroke, and lesion site. The same outcome measurements will be conducted with control participants.

After completion of the project, these sites can consider the implementation of the intervention.

All involved sites work frequently with patients with stroke.

3.2. Project management The project will be led by Hammel Neurocenter (RHN) and University College Nord (UCN). Project phases and studies see Timeline Figure 1.

A. Research lead RHN: a university hospital part of the Department of Clinical Medicine at Aarhus University. On-site is a multidisciplinary research unit with a broad array of methodological competencies. The affiliated Center for post-graduate Education at RHN offers a broad range of post-graduate courses attracting 3200 professionals each year.

UCN: provides higher education and performs research, development, and innovation activities within physiotherapy and other health professions.

Neuroenhed Nord: hosts the Center of Neurotechnology and Rehabilitation, Ålborg University.

B. Project group The steering group will consist of PI Iris Brunner, PT, PhD, associate professor Aarhus University, head of physiotherapy research at RHN; Co-PI Gunhild Mo Hansen, neurological PT, PhD, adjunct lecturer at Fysioterapeutuddannelsen, UCN; Helle Rovsing Jørgensen, MSc, Neuroenhed Nord, Allan Riis, PT, PhD, Research & Development Coordinator at Fysioterapeutuddannelsen, UCN, representatives of the participating municipalities Aalborg, Thisted, Jammerbugt, Skive, Vejle, Favrskov and the participating hospitals Svendborg Neurorehabilitering OUH, and NeuroCentret, Copenhagen.

C. Research assistants Research assistants have crucial functions in conducting all practical aspects regarding recruitment, assessments, delivering follow-up phone calls, and coaching patients. The number of research assistants is only indicative, the tasks can be shared by more people.

3.3. The intervention-ActForStroke Part one High-intensity gait training HIGT is based on substantial amounts of stepping practice at 70-85 % maximum heart rate. Converging data over the past two decades indicate that substantial amounts of stepping practice can improve walking function after stroke without compromising balance or other aspects of gait (14, 19, 20). An algorithm for individual progress has been suggested (21). Therefore, HIGT constitutes a major step towards personalized rehabilitation.

The intervention in practice: Participants in the intervention group will receive 4-5 (at the hospital) or 3 (in municipalty rehabilitation) sessions of HIGT for at least 2 weeks and a maximum of 4 weeks. HIGT will be provided instead of the other physiotherapy interventions such as balance, trunk control, etc.

Part two Facilitating activity Continuous physical activity is crucial for maintaining function and secondary prevention of negative consequences after the most intensive rehabilitation is completed. Research has shown that facilitating techniques, such as motivational interviewing can be effective in encouraging physical activity. Likewise, it has been documented that activity monitoring increases physical activity in adults.

The intervention in practice: Participants in the intervention group will after having participated in HIGT receive coaching based on the Motivational Interviewing counselling approach via phone or video call once a month, up to one year post-stroke. The interviewer will, based on the individual's life situation, together with the individual and their caregivers identify suitable goals for physical activity. Key elements for maintaining physical activity are self-efficacy, motivation, and social support. Consequently, the research staff will try to team up participants with each other, also virtually.

During this period, participants will be monitored with research accelerometers on 3 different occasions for 3 days and will also receive feedback via an app connected to the sensors. Moreover, participants in the intervention group will be encouraged to use their own step counters, e.g., on their smartphones or smartwatches.

Control patients Participants at the control sites will receive the usual type of rehabilitation offered at these sites, including standard gait training. The participants will undergo the same testing procedures and activity monitoring. The participants are free to use any personal monitoring devices, e.g., smartphones or smartwatches.

ELIGIBILITY:
Inclusion Criteria:

* ≥18 years
* stroke within the last 6 months
* able to give informed consent according to the neurorehabilitation team's evaluation and/or cognitive testing
* receiving rehabilitation for post-stroke functional impairments.

Exclusion Criteria:

* Use of bracing or instrumentation (e.g. ventilator) that limits walking independence in walking outdoors and on stairs
* Functional Ambulation Category (FAC) at admission = 5 (independent ambulator on all surfaces)
* uncontrolled cardiopulmonary, metabolic, infectious or psychiatric disorders
* any disorder that prevented walking > 50 meters prior to injury

Min Age: 18 Years | Sex: All | Healthy Volunteers: No
Age Groups: Adult, Older Adult
Enrollment: 50 (Estimated)
Dates: Start 2025-01-01 (Estimated); Primary Completion 2026-07-31 (Estimated); Study Completion 2026-12-31 (Estimated)

PRIMARY OUTCOMES:
Physical activity | From baseline up to 12 months after stroke, 4 assessments will be conducted at inclusion to the study, 2 weeks after inclusion, 6 months and 12 months after stroke.
  The main outcome measure will be the average number of non-sedentary minutes per day measured during 3 days of sensor measurements.
  The SENS motion® wearable sensor will be used to monitor physical activity during 3 days. The SENS motion® registers acceleration on x,y,z axes.

SECONDARY OUTCOMES:
10m walk test | Two assessments: At inclusion to the study, 2 weeks after inclusion.
  Gait assessment
Timed-up-and-go | Two assessments: At inclusion to the study, 2 weeks after inclusion.
  Gait and balance assessment
6 minutes walk test | Two assessments: At inclusion to the study, 2 weeks after inclusion.
  Gait assessment
Sit-to-stand test | Two assessments: At inclusion to the study, 2 weeks after inclusion.
  Assessment of leg strength, describes how many times person can get up from a chair in 1 minute.
Five-level EQ5d (EQ5D) (there is no full name) | Four assessments up to 12 months after stroke: At inclusion, after two weeks, 6 months and 12 months after stroke.
  Quality of life, generic, S The scale ranges from -0.59 to 1 (best)
Stroke Specific Quality of Life (SSQL) | 6 and 12 months after stroke
  Stroke Specific Quality of Life assesses quality of life after stroke. A scale from 12 to 60 (best).
Care giver burden scale | 6 and 12 months after stroke
  Self-reported care giver burden, from 22 (best) to 88 (worst)
Intensity of physical activity | Four measurements up to 12 months after stroke, at inclusion, 2 weeks after inclusion, 6 and 12 months after stroke
  The SENS motion® activity sensor and software will be used to categorize minutes of low, moderate, and high intensity activity during the 3 days of monitoring.
Steps per day | Four assessments up to 12 months after stroke: At inclusion, after two weeks, 6 months and 12 months after stroke.
  The average number of steps per day. SENS motion® activity sensor will be used to monitor steps per day during a 3-day period.

CONTACTS AND LOCATIONS:
Overall Officials: Iris C. Brunner, Phd, Study Director — Aarhus University, Hammel Neurocenter; Gunhild M. Hansen, PhD, Principal Investigator — University College Nord, Aalborg, Denmark
Locations (10):
- Denmark (10):
  - Genoptræning Aalborg Municipality, Aalborg, Denmark
  - Neuroenhed Nord Brønderslev, Brønderslev, Denmark
  - Neurocentet København, Copenhagen, Denmark
  - Hammel Neurocenter and University Research Clinic, Denmark, Hammel, Denmark
  - Favrskov Municipality, Hammel, Denmark
  - Jammerbugt Municipality Neuroteam, Jammerbugt, Denmark
  - Skive Sundhedsafdeling, Skive, Denmark
  - Svendborg Neurorehabilitation, Svendborg, Denmark
  - Thisted Municipality, Thisted, Denmark
  - Vejle Municipality, Vejle, Denmark

IPD SHARING:
Plan to Share IPD: Undecided
Data can be shared as soon as they are totally anonymized.